CLINICAL TRIAL: NCT04340921
Title: The Role of Adaptive Immunity in COVID-19 Associated Myocardial Injury
Status: Withdrawn | Type: Observational
Why Stopped: Failure to recruit
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 282289
Record Dates: First submitted 2020-04-03; First posted 2020-04-10 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Disease Acute; Cardiomyopathies; COVID
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1. COVID-19+ (n=120): COVID-19 positive without evidence of myocardial injury (n=120). Inclusion criteria: All adult (age≥18 but <100 years of age) inpatients with confirmed COVID-19 infection.
  Exclusion criteria: No biochemical evidence of acute myocardial injury (serum troponin>99th centile within previous 48-hour period).
  Interventions: Biological: COVID-19 exposure
- 2. COVID-19+ Myocardial injury+ (n=20): COVID-19 positive with myocarditis (n=20). Inclusion criteria: All adult (age≥18 but <100 years of age) inpatients with confirmed COVID-19 infection and clinically suspected or confirmed myocarditis including evidence of acute myocardial injury (troponin >99th centile within the previous 48-hour period) at the time of recruitment.
  Exclusion criteria: significant chronic kidney disease (eGFR ≤30 or dialysis-dependent) or septic shock at the time of initial assessment. We will also exclude patients with a diagnosis of chronic heart muscle disease and those with known significant chronic or acute obstructive coronary disease.
  Interventions: Biological: COVID-19 exposure
- 3. COVID-19+ Complication+ (estimated 10-25%): Inclusion criteria: Participants form Groups 1 and 2 in whom a prespecified complication ocurs will be included in a derived Group3.
  Interventions: Biological: COVID-19 exposure

INTERVENTIONS:
Biological: COVID-19 exposure — Observation only

SUMMARY:
COVID-19 is associated with complications including ARDS and myocardial injury, which informs prognosis and patient outcome. The laboratory plans to perform immunophenotyping of peripheral T-cells in patients with COVID-19 and complications (ARDS, ITU admission, myocardial injury) and map this against clinical patient outcomes. The aim is to determine if there is a specific T-cell immunophenotype associated with COVID-19 and/or complications, which can be used to inform prognosis and potential therapies.

DETAILED DESCRIPTION:
Infection with the novel coronavirus COVID-19 is designated a pandemic by the World Health Organisation (WHO).COVID-19 infection can result in severe lung inflammation which, when present, dominates the clinical course for most patients. However, other organs may also be involved and the cardiovascular (CV) system appears to have complex interactions with COVID-19. Published reports suggest evidence of heart muscle damage in 20-40% of hospitalised cases presenting as cardiac chest pain, heart failure, abnormal heart rhythms and cardiac death.

Many affected were previously well, but approximately half of those admitted to hospital COVID-19 have other medical problems, increasing in those requiring ITU admission or those that died. Patients with pre-existing CV conditions have some of the worst outcomes. Although pre-existing disorders reduce an individual's capacity to withstand severe illness, it is also likely that CV diseases may increase the risk of developing complicated COVID-19 disease. Our hypothesis is that immunological abnormalities acquired as a consequence of pre-existing disorders is responsible for this.

A question central to potential therapeutic options is the extent to which COVID-19 related myocardial injury results from viral replication (cytopathic), is immune mediated or is due to other mechanisms. Given that rapid onset cardiac injury can occur at 7-14 days after onset of COVID symptoms we propose to evaluate the contribution of adaptive T-cell mediated immunity in patients with and without myocardial injury. If successful, we may be able to identify treatments that suppress discrete components of the immune system to prevent myocardial damage without depressing protective immune function.

ELIGIBILITY:
Group 1: COVID-19 positive without evidence of myocardial injury (n=120). Inclusion criteria: All adult (age≥18 but <100 years of age) inpatients with confirmed COVID-19 infection. Exclusion criteria: No biochemical evidence of acute myocardial injury (serum troponin>99th centile within previous 48-hour period)

Group 2: COVID-19 positive with myocarditis (n=20). Inclusion criteria: All adult (age≥18 but <100 years of age) inpatients with confirmed COVID-19 infection and clinically suspected or confirmed myocarditis including evidence of acute myocardial injury (troponin >99th centile within the previous 48-hour period) at the time of recruitment.

Exclusion criteria: significant chronic kidney disease (eGFR ≤30 or dialysis-dependent) or septic shock at the time of initial assessment. We will also exclude patients with a diagnosis of chronic heart muscle disease and those with known significant chronic or acute obstructive coronary disease.

Group 3: Group 1 and 2 study participants with a complicated course (estimated 14-35 patients).

Inclusion criteria: Participants form Groups 1 and 2 in whom a prespecified complication ocurs will be included in a derived Group3.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years old admitted to the Barts NHS Trust who have a diagnosis of COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
T-cell immunophenotype | 12 months from enrollment
  T-cell immunophenotype

SECONDARY OUTCOMES:
Mortality | 12 months from enrolment
  death, survival to discharge
ITU admission | 12 months from enrolment
  Admission to the intensive care
Myocardial injury | 12 months from enrolment
  Defined by troponin rise to >99th centile

CONTACTS AND LOCATIONS:
Overall Officials: Sam (Saidi) Mohiddin, MD, Principal Investigator — Barts & The London NHS Trust; Federica Marelli-Berg, PhD, Study Chair — Queen Mary University of London
Locations (1):
- Barts Health Nhs Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared from this project.

REFERENCES:
- [Background] Gurwitz D. Angiotensin receptor blockers as tentative SARS-CoV-2 therapeutics. Drug Dev Res. 2020 Aug;81(5):537-540. doi: 10.1002/ddr.21656. Epub 2020 Mar 4. PMID 32129518
- [Background] Ramchand J, Patel SK, Srivastava PM, Farouque O, Burrell LM. Elevated plasma angiotensin converting enzyme 2 activity is an independent predictor of major adverse cardiac events in patients with obstructive coronary artery disease. PLoS One. 2018 Jun 13;13(6):e0198144. doi: 10.1371/journal.pone.0198144. eCollection 2018. PMID 29897923
- [Background] Cooper LT Jr. Myocarditis. N Engl J Med. 2009 Apr 9;360(15):1526-38. doi: 10.1056/NEJMra0800028. PMID 19357408
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Result] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Result] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Result] Komarowska I, Coe D, Wang G, Haas R, Mauro C, Kishore M, Cooper D, Nadkarni S, Fu H, Steinbruchel DA, Pitzalis C, Anderson G, Bucy P, Lombardi G, Breckenridge R, Marelli-Berg FM. Hepatocyte Growth Factor Receptor c-Met Instructs T Cell Cardiotropism and Promotes T Cell Migration to the Heart via Autocrine Chemokine Release. Immunity. 2015 Jun 16;42(6):1087-99. doi: 10.1016/j.immuni.2015.05.014. Epub 2015 Jun 9. PMID 26070483
- [Derived] Bajaj R, Sinclair HC, Patel K, Low B, Pericao A, Manisty C, Guttmann O, Zemrak F, Miller O, Longhi P, Proudfoot A, Lams B, Agarwal S, Marelli-Berg FM, Tiberi S, Cutino-Moguel T, Carr-White G, Mohiddin SA. Delayed-onset myocarditis following COVID-19. Lancet Respir Med. 2021 Apr;9(4):e32-e34. doi: 10.1016/S2213-2600(21)00085-0. Epub 2021 Feb 19. No abstract available. PMID 33617781